CLINICAL TRIAL: NCT02448550
Title: Comparison of Unfractionated Heparin and Bivalirudin for Percutaneous Coronary Intervention for Stable Angina, Unstable Angina, and Non-ST Segment Elevation Myocardial Infarction
Brief Title: Comparison of Anticoagulation for All-comers Undergoing Percutaneous Coronary Revascularization Trial
Acronym: CALIFORNIA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KP-RRC-CE1
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Percutaneous Coronary Intervention
MeSH Terms: interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bivalirudin (Experimental): Bivalirudin will be used for PCI with bailout glycoprotein 2b3a inhibitor use permitted.
  Interventions: Drug: Bivalirudin
- unfractionated heparin (Active Comparator): Unfractionated heparin will be used for PCI with bailout glycoprotein 2b3a inhibitor use permitted.
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Bivalirudin
  Arms: bivalirudin
Drug: Unfractionated heparin
  Arms: unfractionated heparin

SUMMARY:
The purpose of this trial is to determine whether bivalirudin is non-inferior to unfractionated heparin in patients with stable angina, unstable angina, or non-ST segment elevation myocardial infarction undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing PCI for stable angina, unstable angina, or non-ST segment elevation myocardial infarction.
2. Age 18 years or older.

Exclusion Criteria:

1. Inability to obtain consent
2. Emergency cardiac catheterization for ST-segment elevation myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05-06 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Net adverse clinical events (composite of efficacy and safety [bleeding] endpoints) | 30-days

SECONDARY OUTCOMES:
all cause mortality, myocardial infarction, or unplanned revascularization for ischemia | 30-days
Bleeding Academic Research Consortium grade III or V bleeding events | 30-days

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Los Angeles Medical Center, Los Angeles, California, United States